CLINICAL TRIAL: NCT00259779
Title: A Randomised, Double Blind, Double Dummy, Multicentre Phase III Study Comparing the Efficacy of Budesonide/Formoterol (Symbicort® Forte Turbuhaler®) and Oral Prednisolone + Formoterol (Oxis® Turbuhaler) During Two Weeks, in COPD Patients With an Acute Exacerbation, Followed by Twelve Weeks Open Follow up Period With Budesonide/Formoterol (Symbicort Forte Turbuhaler)
Brief Title: Comparison Between Symbicort® and Prednisolone in COPD
Acronym: SPACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5892L00002; Eudra CT 2005-001090-10; SPACE
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Prednisolone

INTERVENTIONS:
Drug: budesonide/formoterol
  Other Names: Symbicort
Drug: Prednisolone

SUMMARY:
To assess if Symbicort forte Turbuhaler (during two weeks) is as effective as an oral course of prednisolone + Oxis Turbuhaler (during two weeks) for the treatment of an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic obstructive pulmonary disease and an acute exacerbation
* After the acute treatment a simple pulmonary function test shows a value of 30%-60% of the predicted normal value.
* Patients, who, based on the clinical examination after the initial acute treatment, are candidates for a course of oral steroids for the treatment of acute symptoms due to chronic obstructive pulmonary disease

Exclusion Criteria:

* Diagnosis/history of asthma
* Oxygen uptake (saturation) is <92% after the initial acute treatment
* A requirement for regular use of oxygen therapy
* Regular treatment with any inhaled steroid >1 000 µg/day at study entry

Additional inclusion and exclusion criteria will be evaluated by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in one second (FEV1)

SECONDARY OUTCOMES:
Number of patients with treatment failures
Time to first exacerbation
Number of patients developing an exacerbation
Diary cards
Quality of Life
- Adverse Events (AEs)
Serious Adverse Events (SAEs) and Discontinuations due to AEs
Variables will be assessed before and over the 2+12 weeks treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (37):
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Ålbæk
  - Research Site, Christiansfeld
  - Research Site, Erfurt
  - Research Site, Nørager
  - Research Site, Oksbøl
  - Research Site, Sæby
- Finland (4):
  - Research Site, Ekenäs
  - Research Site, Jakobstad
  - Research Site, Lohja
  - Research Site, Porvoo
- Germany (3):
  - Research Site, Berlin
  - Research Site, Leipzig
  - Research Site, Marburg
- Norway (5):
  - Research Site, Fredrikstad
  - Research Site, Harstad
  - Research Site, Molde
  - Research Site, Oslo
  - Research Site, Straume
- Sweden (18):
  - Research Site, Alingsås
  - Research Site, Åkersberga
  - Research Site, Åtvidaberg
  - Research Site, Borlänge
  - Research Site, Gothenburg
  - Research Site, Höllviken
  - Research Site, Kilafors
  - Research Site, Limhamn
  - Research Site, Lindesberg
  - Research Site, Luleå
  - Research Site, Malmo
  - Research Site, Motala
  - Research Site, Örebro
  - Research Site, Sigtuna
  - Research Site, Stockholm
  - Research Site, Trosa
  - Research Site, Tumba
  - Research Site, Uppsala

REFERENCES:
- [Derived] Stallberg B, Selroos O, Vogelmeier C, Andersson E, Ekstrom T, Larsson K. Budesonide/formoterol as effective as prednisolone plus formoterol in acute exacerbations of COPD. A double-blind, randomised, non-inferiority, parallel-group, multicentre study. Respir Res. 2009 Feb 19;10(1):11. doi: 10.1186/1465-9921-10-11. PMID 19228428